CLINICAL TRIAL: NCT07081113
Title: Comparative Effects of Cyriax Mobilization and Muscle Energy Techniques on Functional Recovery Following Fixation of Distal Radius Fractures
Brief Title: Study Comparing Cyriax Mobilization and Muscle Energy Techniques for Improving Arm Function in People Recovering From Surgery for Distal Radius (Wrist) Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cyrixmob
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fracture Fixation; Stiffness of Hand, Not Elsewhere Classified

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Cyriax Mobilization (Experimental): Participants in this group will receive Cyriax Mobilization along with conventional physical therapy and radiocarpal mobilization.
  Interventions: Other: Cyriax Mobilization
- Group B - Muscle Energy Techniques (METs) (Experimental): Participants in this group will receive Muscle Energy Techniques (reciprocal inhibition method) along with conventional physical therapy and radiocarpal mobilization.
  Interventions: Other: Muscle Energy Technique (MET)

INTERVENTIONS:
Other: Cyriax Mobilization — Deep transverse friction massage applied to the wrist and forearm muscles, 3 sessions/week for 4 weeks, along with TENS and hot packs.
  Arms: Group A - Cyriax Mobilization
Other: Muscle Energy Technique (MET) — Isometric contractions performed against therapist resistance to improve range of motion and reduce pain, 3 sessions/week for 4 weeks.
  Arms: Group B - Muscle Energy Techniques (METs)

SUMMARY:
This study aims to compare the effects of Cyriax Mobilization and Muscle Energy Techniques (METs) on functional recovery in patients who have undergone surgical fixation of distal radius fractures. A total of 72 participants between 18 and 40 years old will be randomly assigned to two groups. One group will receive Cyriax Mobilization with conventional therapy, while the other will receive METs with conventional therapy. Treatment will last four weeks with three sessions per week. Researchers will measure grip strength, pain levels, range of motion, and functional ability using standard assessment tools. The goal is to determine which therapy is more effective in improving hand and wrist function after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 40 years Both male and female participants Patients in the post-operative phase (4-5 weeks after distal radius fracture fixation) Patients with post-operative wrist stiffness and limited range of motion

Exclusion Criteria:

Open wounds at the fracture site or other fracture complications History of previous fracture in the same limb Comorbid conditions affecting hand function (e.g., rheumatoid arthritis) Neurological deficits (e.g., wrist drop, carpal tunnel syndrome) Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Baseline, Week 2, Week 4
  Measured using a hand-held dynamometer. The highest value from three trials is recorded in kilograms.